CLINICAL TRIAL: NCT04702256
Title: Induction Therapy for Lupus Nephritis With no Added Oral Steroids: An Open Label Randomised Multicentre Controlled Trial Comparing Oral Corticosteroids Plus Mycophenolate Mofetil (MMF) Versus Obinutuzumab and MMF
Brief Title: Induction Therapy for Lupus Nephritis With no Added Oral Steroids: A Trial Comparing Oral Corticosteroids Plus Mycophenolate Mofetil (MMF) Versus Obinutuzumab and MMF
Acronym: OBILUP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200038; 2020-005835-60 (EudraCT Number); MEDAECNAT-2021-05-0070 (Other: ANSM)
Record Dates: First submitted 2020-11-30; First posted 2021-01-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lupus Nephritis; Systemic Lupus Erythematosus (SLE)
Keywords: lupus nephritis; obinutuzumab; corticosteroids; non-inferiority
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — Prednisone; Mycophenolic Acid; Acetaminophen; dexchlorpheniramine; Premedication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obinutuzumab arm (Experimental): Obinutuzumab administration plus oral mycophenolate mofetil (MMF)
  Interventions: Drug: Obinutuzumab administration; Drug: Administration of methylprednisolone, paracetamol and dexchlorpheniramine
- Corticosteroids arm (Active Comparator): Oral corticosteroids plus MMF
  Interventions: Drug: Administration of Methylprednisolone + Prednisone + Mycophenolate mofetil

INTERVENTIONS:
Drug: Obinutuzumab administration — Obinutuzumab administration by intravenous infusion (IV), IV of methylprednisolone, oral mycophenolate mofetil, no prednisone (or if required for extrarenal manifestation(s): less than 10mg/day at any time, less than 7.5mg/day after 6 months and less than 5mg/day after 9 months).
  Hydroxychloroquine will be strongly recommended for all the patients.
  Other Names: GAZYVARO® administration
  Arms: Obinutuzumab arm
Drug: Administration of Methylprednisolone + Prednisone + Mycophenolate mofetil — IV of methylprednisolone, oral prednisone (according to the PNDS), and oral mycophenolate mofetil.
  Hydroxychloroquine will be strongly recommended for all the patients.
  Other Names: Corticosteroid Series
  Arms: Corticosteroids arm
Drug: Administration of methylprednisolone, paracetamol and dexchlorpheniramine — Prior to infusion of obinutuzumab, patients receiving obinutuzumab will receive premedication including 100 mg of methylprednisolone, paracetamol and dexchlorpheniramine.
  Other Names: Premedication
  Arms: Obinutuzumab arm

SUMMARY:
This is a randomised, open label, controlled non-inferiority phase III multicentre trial.

As primary objective, the study aims to demonstrate that a regimen free of additional oral corticosteroids but with obinutuzumab (and MMF) is non-inferior to a regimen based on oral corticosteroids and MMF in achieving the primary outcome of complete renal response at week 52 without receiving corticosteroids above a prespecified dose.

As secondary objectives, the study aims:

* To compare the efficacy of the treatments in both arms in terms of:

  * partial plus complete renal response at week 52;
  * proteinuria < 0.8g/g at week 52;
  * extrarenal flares;
  * response as defined by a >4 points reduction in SELENA-SLEDAI score at week 52.
* To compare the safety of the treatments in both arms in terms of occurrence of:

  * toxicity of corticosteroids;
  * serious Adverse Events;
  * serious Infectious Episodes;
  * new damage.
* To compare the number of patients with non-adherence to treatment in both arms.
* To estimate the efficiency of obinutuzumab in this indication.

The ancillary studies will allow:

* To implement a biobank (serum, plasma, DNA, cells and urine) and a bank of renal biopsies for studies that will be part of separate research funding bids (patients will be informed that their samples and data may be used for subsequent studies and offered to consent or not).
* To identify which target therapeutic levels of MMF best predicts response with least toxicity (ancillary study).
* To have long term data on renal function and damage.

DETAILED DESCRIPTION:
Preliminary data show that the anti CD20 monoclonal antibody may effectively replace oral corticosteroids in the induction treatment of lupus glomerulonephritis. The concept of avoiding significant use of corticosteroids would mark a step change in the approach to the treatment of lupus nephritis but the efficacy of such a strategy first needs to be confirmed in a randomised controlled study.

The main aim of this study is to demonstrate that patients with lupus nephritis could be treated successfully without using damaging doses of oral corticosteroids.

Eligible patients will be randomised with 1:1 ratio, between interventional group (obinutuzumab, IV methylprednisolone, no or low dose corticosteroids and MMF) and control group (oral prednisone, IV methylprednisolone and MMF), after signed informed consent obtaining. Randomization will be blocked and stratified by level of proteinuria (<1 g/g versus ≥ 1 g/g). Previous 52 centers will participate to the trial.

Study assessments will occur on a standard of care basis at 15 days, 1, 3, 6, 9 and 12 months (and at any flare or according to the wishes of the investigator). Study assessment will include assessment of disease activity, disease- and treatment-related damage, quality of life, and blood and urine tests as standard of care. In addition, a biobank will be sampled at inclusion. Long-term data on damage and renal function will be collected during standard of care (18 months, 2, 5 and 10 years) in patients who consented.

Population involved: Children (14 years and above) and adults with lupus nephritis ISN/RPS class III or IV (A or A/C) ± V with active lesions in at least 10% of the viable glomeruli, AND urine protein-to-creatinine ratio (uPCR) ≥ 0.5 g/g.

Data Analysis

In summary, the primary outcome is complete renal response (CR), initial analysis will be descriptive, using odds ratios and 95% confidence intervals (CIs). Formally CR will be analysed using Intention-To-Treat (ITT) analysis via logistic regression. Following the ITT principle, missing data will be imputed. The model will include the treatment effect, and the factors used for stratification in the randomisation as covariates. Odd ratios and 95% CIs derived from the logistic regression will be provided. The results (comparison between the groups) will be presented as an Odds Ratio (OR) (and a two-sided 95% CI) and the trial will be deemed to have met its objective of non-inferiority if the lower bound of the CI (equivalent to a one-sided 97.5% CI) is above a critical value of 0.45 as described above.

Secondary outcomes will be analysed using analogous models with logistic regression for binary endpoints, Cox regression for time-to-event endpoints and multiple linear regression for continuous endpoints. Where appropriate, repeated measures analyses will also be used. The tests will however be two-sided at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 14-17 years old and adults;
* Active lupus nephritis, as defined by kidney biopsy within the preceding 8 weeks, assessed by the International Society of Nephrology/Renal Pathology Society (ISN/RPS) classification: class III or IV (A or A/C) ± V with active lesions in at least 10% of the viable glomeruli;
* Urine protein-to-creatinine ratio (uPCR) ≥ 0.5 g/g at any time in the 14 days before inclusion;
* No contraindications to the use of IV methylprednisolone, MMF, oral corticosteroids or obinutuzumab;
* Ability to provide informed consent;
* Willingness to use appropriate contraception, as recommended when using MMF.

Exclusion Criteria:

* Severe "critical" SLE flare defined as any SLE manifestation requiring more immunosuppression than allowed in the protocol, in the physician's opinion;
* Patients who cannot be prescribed 10 mg prednisone corticosteroids "only", after inclusion according to the physician's opinion;
* Pregnant and breastfeeding woman;
* Prior use within 6 months of inclusion of therapeutic monoclonal antibody and/or B- or T cell modulating 'biologic' except belimumab that can be used up to 7 days before inclusion;
* Obsolescence of >60% of the glomeruli or tubulointerstitial scarring of >60%;
* CKD stage 4 or stage 5 defined as eGFR <30 ml/min/1.73 m2 according to CKD-EPI (to be differentiated from acute renal injury);
* Active infections, including but not limited to human immunodeficiency virus (HIV), hepatitis B in the absence of a specific therapy, hepatitis C or tuberculosis;
* Receipt of a live-attenuated vaccine in the 4 weeks prior to study enrolment;
* History of cervical dysplasia CIN Grade III, cervical high-risk human papillomavirus or abnormal cervical cytology other than abnormal squamous cells of undetermined significance (ASCUS) in the past 3 years in female patients. However, the patient will be eligible in the following conditions: follow-up HPV test is negative or cervical abnormality was effectively treated >1 year ago.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Complete renal response (CR) | at week 52
  CR at week 52 without receiving corticosteroids above a prespecified dose.
  CR at week 52 is defined as:
  * Urine PCR (protein to creatinine ratio) < 0.5 g/g in a spot urine AND:
  * eGFR (estimated glomerular filtration rate using CKD-epi) ≥ 60 ml/min, or if < 60 ml/min at screening, no decline >20% compared to screening/randomisation (whichever worse)
  * AND:
    * In the obinutuzumab arm: with no steroids or without receiving oral corticosteroids > 10 mg/day within the first 6 month, and then, without receiving oral corticosteroids > 7.5 mg/day between 6 and 9 months and > 5 mg/day between 9 and 12 months for SLE indication (according to the French PNDS for SLE after 6 months).
    * In the steroid arm: without receiving corticosteroids above the prescribed taper (according to the French PNDS for SLE, see Appendix A), including without receiving oral corticosteroids > 7.5 mg/day between 6 and 9 months and > 5 mg/day between 9 and 12 months for SLE indication (according to the French
Proteinuria measurement | at baseline
  Proteinuria measurement: the proteinuria/creatinuria ratio will be assessed on a 24-hour urine collection.
Proteinuria measurement | at week 52
  Proteinuria measurement: the proteinuria/creatinuria ratio will be assessed on a 24-hour urine collection.

SECONDARY OUTCOMES:
Efficacy: partial renal response (PR) | at baseline and at week 52
  Partial renal response (PR) will be defined as:
  * 50% improvement in uPCR;
  * AND: uPCR between 0.5 and 3 g/g;
  * AND: no more than a 20% decrease of eGFR from the baseline value (using CKD-epi).
Efficacy: complete renal response | at baseline and at week 52
  Complete renal response: same as in primary outcome.
Efficacy: proteinuria measurement | at baseline and at week 52
  Proteinuria measurement (same as in primary outcome): the proteinuria/creatinuria ratio will be assessed on a 24-hour urine collection.
Efficacy: extrarenal flare | at baseline and at week 52
  Extrarenal flare will be defined according to the SELENA-SLEDAI flare index.
Efficacy: changes in the SELENA-SLEDAI score | at baseline and at week 52
  Changes in the SELENA-SLEDAI score will be measured between inclusion and week 52.
Safety: toxicity of corticosteroids measurement | at inclusion, at Month 6 and Month 12
  The toxicity of corticosteroids will be measured by the Glucocorticoid Toxicity Index (GTI).
  This Composite GTI will be scored (will not be measured separately) with BMI, glucose tolerance, blood pressure, lipid profile, steroid myopathy, skin, neuropsychiatric and ophthalmological toxicity and infections.
Safety: serious adverse events (SAE) report | through study completion, an average of 10 years
  The number of serious adverse events will be measured per patient according to the CTCAE toxicity grading system for the following adverse events combined: death (all causes), grade 3 or higher infections, hospitalization resulting either from the disease or from a complication due to the study treatment.
Safety: number of serious infectious episodes | through study completion, an average of 10 years
  The number of serious infectious episodes will be measured per patient according to the CTCAE toxicity grading system for the following adverse events combined: death (all causes), grade 3 or higher infections.
Safety: changes in the SLICC/ACR damage index. | at inclusion, at Month 6 and Month 12
  New damage will be assessed by measuring changes in the SLICC/ACR damage index.
Non-adherence to treatment: hydroxychloroquine blood levels | at Month 6 and Month 12
  Non-adherence will be defined by otherwise unexplained HCQ drug level < 200 ng/ml and/or undetectable metabolite, at least once during the follow-up visits.
  Non-adherence to treatment will be assessed with hydroxychloroquine blood levels as routinely done in France.
Non-adherence to treatment: questionnaires MASRI | at Month 6 and Month 12
  Non-adherence to treatment will be assessed using questionnaires MASRI.
Efficiency | at one year
  The 1-year total costs of treatment in both arms will be estimated and the incremental cost effectiveness ratio as the difference in costs divided by the difference in QALys estimated from the EQ 5D self-administered questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie COSTEDOAT-CHALUMEAU, MD, PhD, Principal Investigator — Centre de référence maladies auto-immunes et systémiques rares, Internal medicine, Cochin hospital, APHP; Eric DAUGAS, MD, PhD, Study Director — Nephrology department, Bichat Hospital, APHP, Paris
Locations (1):
- Internal medicine, Cochin hospital, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuse H, Akimoto S, Ito H, Shimazaki J, Ishikawa T. [Clinical observations of Cushing's syndrome]. Nihon Hinyokika Gakkai Zasshi. 1984 Aug;75(8):1280-7. doi: 10.5980/jpnjurol1928.75.8_1280. No abstract available. Japanese. PMID 6513226
- [Background] Wofsy D, Hillson JL, Diamond B. Abatacept for lupus nephritis: alternative definitions of complete response support conflicting conclusions. Arthritis Rheum. 2012 Nov;64(11):3660-5. doi: 10.1002/art.34624. PMID 22806274
- [Background] Dall'Era M, Cisternas MG, Smilek DE, Straub L, Houssiau FA, Cervera R, Rovin BH, Mackay M. Predictors of long-term renal outcome in lupus nephritis trials: lessons learned from the Euro-Lupus Nephritis cohort. Arthritis Rheumatol. 2015 May;67(5):1305-13. doi: 10.1002/art.39026. PMID 25605554
- [Background] Costedoat-Chalumeau N, Houssiau F, Izmirly P, Le Guern V, Navarra S, Jolly M, Ruiz-Irastorza G, Baron G, Hachulla E, Agmon-Levin N, Shoenfeld Y, Dall'Ara F, Buyon J, Deligny C, Cervera R, Lazaro E, Bezanahary H, Leroux G, Morel N, Viallard JF, Pineau C, Galicier L, Van Vollenhoven R, Tincani A, Nguyen H, Gondran G, Zahr N, Pouchot J, Piette JC, Petri M, Isenberg D. A Prospective International Study on Adherence to Treatment in 305 Patients With Flaring SLE: Assessment by Drug Levels and Self-Administered Questionnaires. Clin Pharmacol Ther. 2018 Jun;103(6):1074-1082. doi: 10.1002/cpt.885. Epub 2017 Nov 9. PMID 28925027
- [Background] Costedoat-Chalumeau N, Galicier L, Aumaitre O, Frances C, Le Guern V, Liote F, Smail A, Limal N, Perard L, Desmurs-Clavel H, Boutin du LT, Asli B, Kahn JE, Pourrat J, Sailler L, Ackermann F, Papo T, Sacre K, Fain O, Stirnemann J, Cacoub P, Jallouli M, Leroux G, Cohen-Bittan J, Tanguy ML, Hulot JS, Lechat P, Musset L, Amoura Z, Piette JC; Group PLUS. Hydroxychloroquine in systemic lupus erythematosus: results of a French multicentre controlled trial (PLUS Study). Ann Rheum Dis. 2013 Nov;72(11):1786-92. doi: 10.1136/annrheumdis-2012-202322. Epub 2012 Nov 10. PMID 23144449
- [Background] Costedoat-Chalumeau N, Amoura Z, Hulot JS, Aymard G, Leroux G, Marra D, Lechat P, Piette JC. Very low blood hydroxychloroquine concentration as an objective marker of poor adherence to treatment of systemic lupus erythematosus. Ann Rheum Dis. 2007 Jun;66(6):821-4. doi: 10.1136/ard.2006.067835. Epub 2007 Feb 26. PMID 17324970
- [Background] Costedoat-Chalumeau N, Pouchot J, Guettrot-Imbert G, Le Guern V, Leroux G, Marra D, Morel N, Piette JC. Adherence to treatment in systemic lupus erythematosus patients. Best Pract Res Clin Rheumatol. 2013 Jun;27(3):329-40. doi: 10.1016/j.berh.2013.07.001. PMID 24238690
- [Background] Jolly M, Galicier L, Aumaitre O, Frances C, Le Guern V, Liote F, Smail A, Limal N, Perard L, Desmurs-Clavel H, Boutin DL, Asli B, Kahn JE, Pourrat J, Sailler L, Ackermann F, Papo T, Sacre K, Fain O, Stirnemann J, Cacoub P, Jallouli M, Leroux G, Cohen-Bittan J, Hulot JS, Arora S, Amoura Z, Piette JC, Costedoat-Chalumeau N; PLUS group. Quality of life in systemic lupus erythematosus: description in a cohort of French patients and association with blood hydroxychloroquine levels. Lupus. 2016 Jun;25(7):735-40. doi: 10.1177/0961203315627200. Epub 2016 Feb 13. PMID 26876692
- [Derived] Dossier C, Hogan J. Response to Majeranowski. Pediatr Nephrol. 2021 Jun;36(6):1653. doi: 10.1007/s00467-021-04982-4. Epub 2021 Mar 10. No abstract available. PMID 33693991